CLINICAL TRIAL: NCT04365829
Title: Tolerance for Using Virtual Reality With Subjects Living in Accommodation Establishment for the Elderly Dependent (EHPAD)
Acronym: RAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00377-32
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Anxiety Disorders; Residents of Retirement Home (EHPAD)
Keywords: Residents of Retirement Home (EHPAD); Virtual reality; anxiety disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality (Experimental)
  Interventions: Device: virtual reality headset "Occulus GO"

INTERVENTIONS:
Device: virtual reality headset "Occulus GO" — Use of a virtual reality headset for one week at a frequency of 3 days per week (D1, D3 and D5). During each session (1 hour), the subject will visualize a scene of natural virtual environment (a garden, animals in the wild, a grand Canyon) lasting 7 min using an virtual reality headset "Occulus GO".

SUMMARY:
The main purpose of this study is to assess the tolerance of the virtual environment in the elderly living in a nursing home (EHPAD). It will be evaluated by the cybersickness collection after each session (1 session every other day for a total of 3 sessions).

DETAILED DESCRIPTION:
The purpose of this muliticentric, interventional, uncontrolled study is to assess the tolerance of the virtual environment in the elderly living in a nursing home

subjects who fulfil the inclusion criteria and after signing the informed consent will benefit from three individual virtual reality (VR) sessions.

The sessions will be performed out with one day apart

An assessment of anxiety trait and well-being of each subject will be performed before the first session (D1) and after the third (D3).

An assessment of anxiety as a condition will be performed before and after each session.

Heart rate and blood pressure measurements will be made before, during and after each session.

At the end of each session, an evaluation of cybersickness will be performed. Feedback on the acceptability of the experience will be provided at the end of each session.

Each session will last 1 hour in total: the person will visualize a single scene of virtual reality presenting a natural environment of a duration of 7 minutes preceded by a time of introduction, evaluation and followed by a time dedicated to evaluations and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination (M.M.S.E) scale ≥ 20.
* University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) scale ≥ 12/20.
* Living in Retirment Homes (EHPAD).
* Good understanding of the French language.
* Benefiting from a social security scheme.
* Have read the newsletter and have consented to participate in the study by signing a written consent.

Exclusion Criteria:

* History of epileptic seizures.
* Taking antihypertensive, neuroleptic, tricyclic antidepressants or parkinsonian drugs
* Psychiatric disorders (Schizophrenia, dissociative disorders, borderline states, paranoia).
* Hypertension (unless it is stabilized due to the absence of a change in antihypertensive treatment in the last 3 months and without a notable episode of orthostatic hypotension reported).
* Vestibular or cerebellar syndromes.
* Subjects under legal protection (curatorship, tutorship and safeguard of justice).
* Refusal to participate.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Assess the tolerance of the virtual environment according Simulator sickness questionnaire | 5 days

SECONDARY OUTCOMES:
Assessment of the trait and the state of anxiety according a psychological inventory "State-Trait Anxiety Inventory" scale (STAI-Y) | 5 Days
  The State-Trait Anxiety Inventory (STAI-Y) is a psychological inventory based on a 4-point Likert scale. Higher scores are positively correlated with higher levels of anxiety.
Measuring current mental wellbeing according "World Health Organisation- Five Well-Being" Index (WHO-5) | 5 Days
  The total score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Measuring Heart Rate according the tensiometer | 5 Days
Measuring Blood Pressure according the tensiometer | 5 Days
  both systolic and diastolic blood pressure will be measured
evaluation of the impression on the Virtual Reality (VR) experience, the emotions aroused by it the motivation to renew it according to "Acceptability Questionnaire" | 5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DURON, MD, Study Chair — Geriatric Department, Paul Brousse Hospital
Locations (1):
- Geriatric Department, Paul Brousse Hospital, Villejuif, IIe-de-France, France